CLINICAL TRIAL: NCT07022184
Title: A Personalized Lifestyle Intervention for Depression Symptomatology in General Practice - a Cluster Randomized Multicenter Trial
Brief Title: Lifestyle Intervention for Symptoms of Depression wIth App Support in General Practice
Acronym: LIDIAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ixta Noa (Unknown); Hogeschool van Arnhem en Nijmegen (HAN) (Unknown); Pro Persona Mental Health Care Foundation (Other); Amsterdam UMC (Other); Interactive Studios (Unknown); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-17656; 10930012310037 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-05-22; First posted 2025-06-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Depressive/Anxiety Symptoms; Depressive Disorder
Keywords: Personalized lifestyle intervention; eHealth; Measurement-based care; Depression symptomatology; Cluster randomized trial; General practice; Lifestyle changes; Mental health support; Primary care
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care As Usual (CAU) (No Intervention): The control group, receiving care as usual, will use a version of the Patient Journey App that only displays study questionnaires and sends reminders to complete them at the start of the study, and again at 3 and 6 months. Every 6 weeks, depression symptoms are measured. Patients can view their depression questionnaire results (PHQ-9; Patient Health Questionnaire-9) in a graph within the app. General practitioners and mental health nurses will not have access to the app. At 12 months, all participants will be invited to complete an optional final questionnaire about (cost-)effectiveness to assess the long-term impact of the intervention.
- Personalized Lifestyle Intervention (Experimental): The intervention group will receive the personalized lifestyle intervention (PLI) in addition to care as usual. The PLI consists of the combined use of the Patient Journey App and regular treatment provided by the general practitioner or mental health nurse in general practice. Patients, general practitioners and mental health nurses will have access to the app to monitor patient progress and outcomes (symptoms of depression and anxiety). Study questionnaires will be completed at the start of the study (baseline), and again at 3, 6, and optionally 12 months after enrollment. Every 6 weeks, depression symptoms are measured.
  Interventions: Device: Personalized Lifestyle Intervention

INTERVENTIONS:
Device: Personalized Lifestyle Intervention — The personalized lifestyle intervention (PLI) consists of the combined use of the Patient Journey App (PJA) alongside care provided by the general practitioner or mental health nurse.
  The Patient Journey App integrates four digital health tools within a single smartphone application:
  1. A brief lifestyle questionnaire covering six key areas: mental wellbeing, minimizing harmful substance use, social relationships, healthy eating, sleep, and physical activity.
  2. A personalized summary of the questionnaire results, which supports the formulation of two personal lifestyle goals.
  3. Tailored information and advice about lifestyle, including suggested interventions, based on the patient's personal goals.
  4. Monitoring of depression symptoms over time to support measurement-based care.
  General practitioners and mental health nurses will have access to the app to monitor patient progress and outcomes.
  Other Names: Patient Journey App; Lifestyle App; PLI
  Arms: Personalized Lifestyle Intervention

SUMMARY:
The goal of this clinical trial is to find out whether a smartphone app can help reduce symptoms of depression by supporting healthy lifestyle changes and encouraging self-monitoring in adults who visit their general practitioner with symptoms of depression.

The main questions this study aims to answer are:

Does a personalized lifestyle intervention delivered through the app, in addition to regular care, reduce depression symptoms more effectively than regular care alone? Is this approach more cost-effective than regular care alone?

Researchers will compare patients who use the app alongside their regular care to patients who receive regular care without the app, to see whether the app leads to better outcomes.

Participants who use the app will:

Complete a lifestyle questionnaire focused on six themes: mental wellbeing, use of harmful substances, social relationships, healthy eating, sleep, and physical activity.

Set personal goals based on their results and receive tailored lifestyle advice.

Track their depression symptoms regularly within the app to support ongoing care.

Have follow-up conversations with their general practitioner or mental health nurse to discuss their progress.

Fill out questionnaires about their symptoms and experiences during the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing an episode of symptoms of depression and receiving treatment for this episode from their GP or GP-MHW for less than six months
* Have a smartphone
* Be proficient in Dutch

Exclusion Criteria:

* Severe mental illness (such as psychosis or bipolar disorder)
* Severe alcohol or drug addiction requiring specialized secondary care
* High suicide risk
* moderate to severe cognitive impairment (as determined by the GP)

Patients who visit their GP for depressive symptoms but with a PHQ-9 of <5 at baseline are allowed to use the PLI, but will not be included in the primary analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness of the Personalized Lifestyle Intervention at 6 months after baseline | Baseline to 6 months
  To assess the PLI's cost-effectiveness from a societal perspective, the Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) will be used. The main outcome in the cost-effectiveness analysis is Quality-Adjusted Life-Years (QALYs) based on the EQ-5D-5L, measuring general quality of life.
  Also, additional treatments are measured within the TIC-P, for secondary analysis on additional care.
Change in quality of life using the EQ-5D-5L | Baseline to 6 months
  Change in quality of life will be assessed using the EQ-5D-5L. This tool consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with each rated on a 5-level scale. The EQ-5D-5L also includes a visual analog scale (VAS) to assess overall health. Higher scores indicate better quality of life, while lower scores reflect greater limitations or discomfort. This measure helps track changes in health status and overall quality of life over time.
Change from baseline in the mean depression severity score measured by the PHQ-9 at 6 months after baseline | Baseline to 6 months.
  To evaluate the effectiveness of the PLI on depression symptomatology, general symptoms of depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-reported questionnaire assessing the severity of depression symptomatology. The PHQ-9 is brief, easy to complete, and takes only a few minutes to fill out. The total score ranges from 0 to 27. Scores are interpreted as follows: 0-4 indicates minimal or no depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression. Higher scores suggest more severe symptoms, and professional treatment is recommended as the score increases.

SECONDARY OUTCOMES:
Change in the severity of anxiety symptoms: GAD-7 (Generalized Anxiety Disorder-7) | Baseline to 3 , 6 and 12 months
  To measure the severity of anxiety symptoms, the GAD-7 (Generalized Anxiety Disorder-7) will be used
Changes in quality of life according to the Recovering Quality of Life (ReQol) | Baseline to 3, 6 and 12 months
  Quality of life is measured using the Recovering Quality of Life (ReQol) questionnaire, a patient-reported outcome measure specifically developed for individuals with various mental health conditions. The ReQol provides a total score ranging from 0 to 80, with higher scores reflecting a better quality of life and overall recovery outcome.
Change in use of antidepressants | Baseline to 3 and 6 months
  Use of antidepressants, when started/ended, type, dosage, and at follow-up: inquire about changes.
Change in use of anxiolytics | Baseline to 3 and 6 months
  Use of anxiolytics by self-reported questions about the use of sedatives/sleep medication, when started/ended, frequency of use, type, dosage, and at follow-up: inquire about changes.
Change in lifestyle measures at month 6 | Baseline to 6 months
  Self-constructed questions about the daily lifestyle habits of all participants. The lifestyle components addressed include smoking, alcohol consumption, drug use, sleep duration, adherence to the Dutch Physical Activity Guidelines according to the Dutch National Institute for Public Health and the Environment (RIVM), and nutrition based on the dietary recommendations of the Netherlands Nutrition Centre.
Change in BMI | Baseline to 6 months
  Weight and height will be combined to report BMI (Body Mass Index) in kg/m^2.
Change in lifestyle satisfaction measures at month 6 (intervention arm) | Baseline (intervention only) and 6 months (both groups)
  In the intervention group, self-constructed questions about lifestyle are used to measure a patient's satisfaction with specific lifestyle components on a scale from 0 to 10, where 10 indicates the highest level of satisfaction. The lifestyle components include mental wellbeing, minimizing harmful substances, social relationships, healthy eating, sleep, and physical activity. It is possible that someone smokes but is currently satisfied with this and does not wish to make any changes. The intervention is not intended to impose certain behaviors but rather to address the lifestyle components that the individual is willing and motivated to improve, with the ultimate goal of reducing depressive symptoms. These questions collectively provide an overview that the healthcare provider and patient can use together to set achievable goals. In the control group, this questionnaire will only be completed at month 6 of the study.
Patient satisfaction: CQi (Consumer Quality Index) | At 6 months
  The Consumer Quality Index (CQI) is a 16-item questionnaire that evaluates patient experiences and satisfaction across various dimensions, such as communication, access to care, and treatment outcomes. The CQI helps healthcare providers track patient experiences and identify opportunities for enhancing care. It has a 5 point scale. The last item is a scoring item for overall treatment satisfaction. Higher scores indicate better satisfaction, while lower scores highlight areas for improvement.
Change in patient-doctor relationship: PDRQ-9 | Baseline to 6 months
  The Patient-Doctor-Relationship Questionnaire (PDRQ-9) is a patient-reported outcome measure used to assess the quality of the therapeutic relationship between patients and their healthcare providers, such as general practitioners (GPs) or mental health nurses (GP-MHNs). The questionnaire evaluates key aspects of the patient-provider interaction, helping to capture the perceived level of trust, support, and communication. The score ranges from 9 to 45, higher score indicating a more positive relationship according to the patient.
Change in social support: SSL12 (Social Support List-12) | Baseline to 6 months
  Social support will be measured using the SSL12 (Social Support List-12) questionnaire. This validated tool assesses perceived social support across various domains, such as emotional, practical, and informational support. Higher scores indicate greater perceived social support, while lower scores suggest limited support. The SSL12 helps evaluate the level of social assistance individuals feel they receive and can track changes in social support over time.
PHQ-9 at 3 and 12 months | Baseline to 6 weeks, 3 months and 12 months
  Secondary analysis of PHQ-9 outcomes. To evaluate the effectiveness of the PLI on depression symptomatology, general symptoms of depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9) every 6 weeks. The PHQ-9 is a 9-item self-reported questionnaire assessing the severity of depression symptomatology. The PHQ-9 is brief, easy to complete, and takes only a few minutes to fill out. The total score ranges from 0 to 27. Scores are interpreted as follows: 0-4 indicates minimal or no depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression. Higher scores suggest more severe symptoms, and professional treatment is recommended as the score increases.
Cost-effectiveness at 3 months and at 12 months | baseline to 3 and 12 months
  To assess the PLI's cost-effectiveness from a societal perspective, the Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) will be used. The main outcome in the cost-effectiveness analysis is Quality-Adjusted Life-Years (QALYs) based on the EQ-5D-5L, measuring general quality of life. At 3 and 12 months, an incremental analysis is done in addition to the cost-effectiveness at 6 months

OTHER OUTCOMES:
Socio-demographics at baseline | At baseline
  Baseline demographics include gender, age, education level, employment status and ethnicity.
Threatening Experiences: LTE | At enrollment and at 6 months
  The List of Threatening Experiences (LTE, developed bij Brugha) measures the occurrence of 12 major categories of stressful life events (did you experience this: No, yes in the last 6 months, yes longer ago) The Dutch translation includes an additional thirteenth question: "Did you experience any other major severe negative events (yes/no)? If yes, briefly describe what happened?" The questionnaire is offered at baseline, and at 6 months a shorter version (did you experience this in the last 6 months?).
  Item scores are summed to derive a total score. Higher score indicates more threatening experiences.
History of depression and previous psychological treatment | At baseline
  History of depression and previous psychological treatment are assessed through self-reported questions. These include the number of previous depressive episodes treated, the number of hospitalizations for depression in a psychiatric hospital or mental health institution, age of onset, duration of the current episode (when it began), family history of depression, and any previous psychological treatment or psychotherapy.
Chronic diseases: TIC-P | At baseline
  Chronic diseases will be evaluated using questions of the TIC-P questionnaire e.g., health status, lung diseases, heart diseases, blood vessels, diabetes, stroke, joint degeneration, rheumatism, cancer, high blood pressure, and other diseases.
Psychiatric comorbidities: LIDAS items (LIfetime Depression Assessment Self-report), adjusted. | Baseline to month 6
  This questionnaire comprises questions about psychiatric diagnoses and treatment (in the last 6 months , ever or never), other than depression.
Meta-data Patient Journey App during study | At 6 and 12 months
  Meta-data in the Patient Journey App will be tracked and analyzed. Meta-data includes application usage data such as the frequency of app openings, the number of times patients access information, and which features or sections are most frequently used or viewed.
Acceptability and usability of the app: modified MAUQ (intervention arm) | At 6 months (intervention arm only).
  The mHealth App Usability Questionnaire (MAUQ) is a 21-item survey scored on a 7 point likert scale from 1 (disagree) to 7 (agree) with higher scores indicative of higher usability. For this study, the subscales MAUQ-E (8 items on Ease of use and satisfaction) and MAUQ-U (7 items on Usefulness) will be used.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Amsterdam UMC, Amsterdam, North Holland
  - UMC Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study website LIDIAS — https://www.radboudumc.nl/lopende-onderzoeken/lidias